CLINICAL TRIAL: NCT06543524
Title: Survival and nEonatal outComes of veRy Low Birth wEight Infants in Türkiye: Turkish Neonatal Society SECRETS-TR Study
Acronym: TNS-SECRETS
Status: Completed | Type: Observational
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Collaborators: Turkish Neonatal Society (Other)
Responsible Party: Principal Investigator, Merih CETINKAYA, Professor, MD, PhD, Başakşehir Çam & Sakura City Hospital
Other Study IDs: TNS001
Record Dates: First submitted 2024-07-28; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Morbidity;Infant
Keywords: prematurity,; very low birth weight infant; outcomes; mortality; morbidity
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Care of premature infants — No intervention was performed

SUMMARY:
The aim of this multi-center study was to evaluate the mortality rate and early neonatal outcomes of very low birth weight (VLBW) infants hospitalized in neonatal intensive care units (NICUs) in Türkiye. It was promoted by the Turkish Neonatology Society (TNS) and research was approved by the Cam and Sakura City Hospital Ethical Committee.

It was conducted between 28 April 2021 and 02 January 2023 and written informed consents from the families of included patients were obtained.

A total of 74 level III and IV NICUs participated to the study. All the centers had an oppurtunity to follow-up these high risk premature infants in terms of their medical staff, equipment and other neonatology sources.

The inclusion criteria consisted of preterm infants with birth weight (BW)≤1500 grams and with gestational age (GA) of 24 0/7 weeks to 31 6/7 weeks, all inborn and outborn infants admitted to NICU within the first 24 hours of life and approval of parental consent.The survival status, maternal, perinatal and neonatal characteristics, risk factors and early neonatal outcomes of all infants were recorded.

DETAILED DESCRIPTION:
The study includes the selected cohort of approximately 3000 very low birth weight preterm infants born in one year period in Turkey in level III/IV neonatal intensive care units (NICUs). Detailed information on antenatal (growth, infection), natal (neonatal resuscitation, non-invasive/invasive ventilation and surfactant administration in the delivery room) and postnatal clinical course in NICUs (ventilatory support, circulation, intestinal and cranial event status,growth, exitus) were recorded. The mortality and overall spesific morbidities of the study population will be evaluated. Also, subgroup analysis for extremely low birth weight infants, micropremies, gray zone infants (22 to 24 weeks of gestational age) will also be performed for local data of Turkey and will be used for development of local guidelines and improvements in the care of preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants with BW≤1500 grams and with gestational age (GA) of 24 0/7 weeks to 31 6/7 weeks,
* All inborn and outborn infants admitted to NICU within the first 24 hours of life
* Presence of parental consent

Exclusion Criteria:

* The larger infants than inclusion criteria,
* Infants who died in the delivery room,
* Infants admitted to NICU after first 24 hours of life,
* Infants with major congenital/chromosomal abnormalities
* Refusal of parental consent

Ages: 60 Minutes to 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Very low birth weight preterm infants with BW≤1500 grams and with gestational age (GA) of 24 0/7 weeks to 31 6/7 weeks and admitted to NICU within the first 24 hours of life
Sampling Method: Probability Sample
Enrollment: 3150 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
mortality rate | during hospitalization period, with an average of 6 months.
  mortality rate of infants participated to the study
rate of prematurity-related morbidities | during hospitalization period or at the time of discharge whichever came first, assessed through study completion, an average of 6 months
  rates of prematurity-related morbidities in infants participated to the study

SECONDARY OUTCOMES:
Duration of hospitalization | at the time of discharge of the Neonatal Intensive Care Unit (NICU), an average of 1 year.
  Length of hospitalization as day

CONTACTS AND LOCATIONS:
Overall Officials: Merih Cetinkaya, Principal Investigator — Başakşehir Çam & Sakura City Hospital
Locations (1):
- BasaksehirCamSakuraSehirH, Istanbul, Please Select, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No